CLINICAL TRIAL: NCT02305615
Title: Hungarian Multicenter Non-Interventional Study of Continued Avastin (Bevacizumab) Plus Chemotherapy Until First Progression Following Induction Treatment With Chemotherapy Doublet Plus Avastin in First Line Treatment of Patients With Metastatic Colorectal Carcinoma
Brief Title: An Observational Study of Continued Bevacizumab Plus Chemotherapy Until First Progression in Participants With Metastatic Colorectal Cancer (CRC)
Acronym: AVACONT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29425
Record Dates: First submitted 2014-11-28; First posted 2014-12-02 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants with CRC: This is an observational study; thus, no intervention or treatment is required by the protocol. During the study, the treatment will be determined according to the treating physician decision. Eligible participants will be observed for safety and efficacy of continued bevacizumab plus fluoropyrimidine-based doublet chemotherapy treatment in routine clinical practice for 1 year.
  Interventions: Other: Bevacizumab; Combination Product: Chemotherapy

INTERVENTIONS:
Other: Bevacizumab — Bevacizumab at a dose and schedule according to approved label and SmPC. The recommended dose of bevacizumab, administered as an intravenous infusion, is either 5 milligrams per kilogram (mg/kg) or 10 mg/kg of body weight given once every 2 weeks or 7.5 mg/kg or 15 mg/kg of body weight given once every 3 weeks. Bevacizumab is always used in combination with chemotherapy for the treatment of participants with metastatic CRC. It is recommended that treatment be continued until progression of the underlying disease or until unacceptable toxicity.
  Other Names: Avastin
Combination Product: Chemotherapy — Fluoropyrimidine-based doublet chemotherapy (5-Fluorouracil [5-FU] or capecitabine plus oxaliplatin or irinotecan) as first-line treatment; and continued fluoropyrimidine treatment with or without treatment modification for oxaliplatin or irinotecan, as per treating physician discretion.

SUMMARY:
This prospective, multicenter, observational study will investigate the effectiveness and safety of bevacizumab in routine clinical practice in participants with metastatic CRC. Participants are to have initiated first-line treatment with fluoropyrimidine-based doublet chemotherapy plus bevacizumab according to the bevacizumab Summary of Product Characteristics (SmPC).

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed CRC with metastatic lesion
* Participants having initiated first-line treatment with fluoropyrimidine-based doublet chemotherapy plus bevacizumab according to bevacizumab SmPC
* Participants who previously received a minimum 9 cycles of 5-FU-based or a minimum 6 cycles of capecitabine-based induction doublet chemotherapy (i.e. 5-FU or capecitabine + oxaliplatin or irinotecan) plus bevacizumab
* Disease evaluation showed stable disease, partial response, or complete response according to RECIST within one month

Exclusion Criteria:

* Contraindication to receive bevacizumab according to the bevacizumab SmPC
* Participants who received more than 10 cycles of 5-FU-based or more than 7 cycles of capecitabine-based induction doublet chemotherapy plus bevacizumab
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with metastatic CRC in first-line setting in Hungary
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2017-12-29 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to the first documented progression or death from any cause, whichever occurs first (maximum up to 36 months)

SECONDARY OUTCOMES:
PFS on First-Line Therapy | From first dose of bevacizumab first-line treatment up to the first documented progression or death from any cause, whichever occurs first (maximum up to 36 months)
Percentage of Participants who were Alive at 1 Year | From enrollment up to death from any cause, maximum up to 1 year
Duration of Bevacizumab Plus Chemotherapy Treatment | From Baseline up to 36 months
Percentage of Participants with Best Overall Response Assessed by Treating Physicians Using Response Evaluation Criteria in Solid Tumors (RECIST) | From Baseline up to 36 months
Percentage of Participants with Reason for Bevacizumab Plus Chemotherapy Treatment Discontinuation | From enrollment to the treatment discontinuation (maximum up to 36 months)
Percentage of Participants with Protocol Defined Baseline Participant and Disease Characteristics | Baseline
  Protocol defined baseline participant and disease characteristics include: gender (male, female); age at enrollment (less than [<] 65 years, greater than or equal to [>/=] 65 years); Eastern Cooperative Oncology Group (ECOG) performance status (0,1, >/=2); primary tumor location (colon, rectum); liver metastasis only (yes, no); number and sites of organs with metastases (less than or equal to [</=] 1, greater than [>] 1); prior adjuvant chemotherapy (yes, no); resection of primary tumor (yes, no); disease stage at the time of diagnosis; disease-free interval between CRC disease diagnosis and diagnosis of metastatic stage; and mutation status (RAS, BRAF) if available.
Percentage of Participants with Adverse Events (AEs) and Serious AEs | From Baseline up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Hungary (22):
  - Szent Margit Hospital, Budapest
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Szent Imre Hospital, Budapest
  - Orszagos Onkologiai Intezet; B Belgyogyaszati Osztaly, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Fövárosi Önkormányzat uzsoki utcai Kórház, Budapest
  - Kenezy Korhaz Rendelointezet, Debrecen
  - Debreceni Egyetem Klinikai Kozpont ; Department of Oncology, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Békés Megyei Pándy Kálmán Kórház; Onkologiai tanszek, Gyula
  - Kaposi Mor Teaching Hospital, Kaposvár
  - Bacs-Kiskun Megyei Korhaz, SZTE AOK Oktato Korhaza, Onkoradiologiai Kozpont, Kecskemét
  - Borsod-Abauj-Zemplen Megyei Korhaz Es Egyetemi Oktato Korhaz; Onkologiai Osztaly, Miskolc
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Pécsi Tudományegyetem Áok; Onkoterapias Intezet, Pécs
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
  - Tolna Megyei Onkormanyzat Balassa Janos Korhaz, Szekszárd
  - Szent Gyorgy Korhaz;Fejer Megyei, Székesfehérvár
  - Markusovszky Hospital, Szombathely
  - Szent Borbala Korhaz, Tatabánya
  - Veszprem Megyei Csolnoky; Ferenc Korhaz, Veszprém
  - Zala megyei Önkormányzat Kórház és Rendelõintézet, Zalaegerszeg